CLINICAL TRIAL: NCT00336596
Title: Transcranial Ultrasound Enhanced Thrombolysis (TRUST)
Brief Title: Ultrasound Enhanced Thrombolytic Therapy of Middle Cerebral Artery Occlusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-031/2004
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Intracranial Embolism; Thrombosis
Keywords: middle cerebral artery occlusion; intracranial embolism and thrombosis; ultrasound enhanced thrombolysis; Patients receiving iv thrombolytic therapy (t-PA)
MeSH Terms: conditions — Intracranial Embolism; Thrombosis; Infarction, Middle Cerebral Artery; Intracranial Embolism and Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: transcranial ultrasound in patients treated with iv t-PA

SUMMARY:
The purpose of the present, randomized, controlled multicenter phase III trial is to investigate the safety and efficacy of continuous 1-hour insonation of occluded middle cerebral artery with 2 MHz TCCS in stroke patients treated with intravenous tissue plasminogen activator (t-PA) within 3 hours after symptom onset.

DETAILED DESCRIPTION:
Thrombolysis with intravenous(iv) tissue plasminogen activator (t-PA) is the only effective and approved therapy for acute ischemic stroke. The most frequent cause of ischemic stroke is thrombosis of the middle cerebral artery (MCA). Preliminary in vitro, animal and human studies suggest that ultrasound accelerates thrombolysis induced by t-PA, and recanalization of acute MCA occlusion due to thrombolysis is an independent predictor of good clinical outcome. Thus, insonation of an occluded MCA through the temporal bone in stroke patients who are treated with iv t-PA might enhance recanalization and improve clinical outcome. The present prospective, randomized, controlled multicenter pilot study will investigate the safety and efficacy of continuous 1-hour insonation of the occluded MCA with 2 MHz transcranial color duplex sonography in patients with ischemic stroke treated with iv t-PA within 3 hours after symptom onset. It is planned to randomize 400 patients in 6 Swiss centers during an enrolment period of 33 months with an individual follow up of 3 months. The study endpoints include safety and efficacy assessments. The primary safety endpoint is to determine the rate of symptomatic intracranial hemorrhage (ICH) in both treatment groups. The primary efficacy endpoint is to determine whether a good functional outcome (modified Rankin scale, mRs, score of 0-2) differs between both treatment groups. Secondary endpoints include (1) asymptomatic ICH occuring during or within the first 24-48 hours after t-PA infusion, (2) early clinical recovery by 10 or more National Institute of Health Stroke Scale (NIHSS) points or dramatic recovery (total NIHSS score of 3 or less) at 24-48 hours after t-PA infusion, (3) mean mRS score at 90 days after t-PA infusion, (4) death occuring during the study period, and (5) recanalization at 24-48 hours after t-PA infusion.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke in the MCA territory according to clinical and cranial computed tomography (CT) or cranial MR imaging (MRI) findings
* patient undergoing iv thrombolysis with t-PA within 3 hours after stroke onset
* Occlusion of sphenoidal (M1) or insular (M2) segment of the MCA at CT (CTA), MR (MRA) or catheter (CA) angiography
* appropriate temporal bony window without echocontrast agents for insonation with TCCS
* full functional independence prior to present stroke (mRS 0-1), use of a cane for walking due to comorbid condition is acceptable
* written informed consent, signed and dated by the subject (or subject's authorized representative, if allowed by local laws) and by the person obtaining the consent, indicating agreement to comply with all protocol-specific procedures

Exclusion Criteria:

* unconsciousness (more than 2 points on item 1a on NIHSS)
* history of intracranial hemorrhage, arteriovenous malformation or aneurysm
* severe cranio-cerebral trauma within the last 3 months
* symptoms of subarachnoidal hemorrhage
* time of symptom onset unclear
* large surgical intervention or trauma within the last 10 days
* expected survival below 90 days after iv t-PA treatment
* severe hepatic disease, esophageal varices, acute pancreatitis
* septic embolism, endocarditis, pericarditis after myocardial infarction
* pregnancy or childbirth within the last 30 days or nursing mothers
* history of hemorrhagic diathesis or coagulopathy
* untreatable increase of arterial blood pressure (>185mmHg systolic, >110mmHg diastolic)
* intracranial hemorrhage, arteriovenous malformations or aneurysm at brain imaging
* thrombocytes <100'000 per microliter
* international normalized ratio (INR)>1.7 or partial thromboplastin time (PTT) prolongated
* serum glucose <2.7mmol/l or >22.2mmol/l
* severe renal insufficiency or other contraindications against CT-contrast agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2006-06; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Symptomatic intracranial hemorrhage (safety)
Functional outcome (efficacy)

SECONDARY OUTCOMES:
Asymptomatic intracranial hemorrhage 24-48 hours after t-PA infusion
Early clinical recovery by 10 or more NIHSS points or dramatic recovery (total NIHSS 3 or less)at 24-48 hours after t-PA infusion
Mean mRS score at 90 days after t-PA infusion
Death occurring during study period
Recanalization at 24-48 hours after t-PA infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ralf W Baumgartner, MD, Study Chair — University Hospital of Zurich, Department of Neurology, Zurich, Switzerland
Locations (6):
- Switzerland (6):
  - Kantonsspital Aarau, Department of Neurology, Aarau
  - University Hospital of Basel, Department of Neurology, Basel
  - University hospital of Bern, Department of Neurology, Bern
  - University Hospital of Geneva, Department of Neurology, Geneva
  - University Hospital of Lausanne, Department of Neurology, Lausanne
  - University Hospital of Zurich, Department of Neurology, Zurich